CLINICAL TRIAL: NCT02077959
Title: Phase I/II Study of Lenalidomide in Combination With Anti-PD-1 Monoclonal Antibody CT-011 in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Lenalidomide and Pidilizumab in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pharmaceutical Companies decision
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: CureTech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-13128; NCI-2014-00385 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; pidilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide, pidilizumab) (Experimental): Patients receive lenalidomide PO daily on days 1-21 and pidilizumab IV over 1-2 hours on day 3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide; Biological: pidilizumab; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Biological: pidilizumab — Given IV
  Other Names: CT-011
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide and pidilizumab and to see how well they work in treating patients with multiple myeloma that has come back (relapsed) or has not responded to treatment (refractory). Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as pidilizumab, can block cancer growth by blocking the ability of cancer to grow and spread. Giving lenalidomide with pidilizumab may work better in treating relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD), safety and efficacy of CT-011 (pidilizumab) in combination with lenalidomide (Revlimid) and assess efficacy in terms of overall response rate in patients with relapse/refractory multiple myeloma (MM).

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study but this phase did not move forward.

Patients receive lenalidomide orally (PO) daily on days 1-21 and pidilizumab intravenously (IV) over 2 hours on day 3. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients have evidence of relapse or refractory disease as defined by International Myeloma Working Group (IMWG) criteria and measurable disease as defined by any of the following:

  * Serum M-protein >= 0.5 g/dl (>= 10 g/l)
  * Urine monoclonal protein >= 200 mg/24h
  * Involved free light chain (FLC) level >= 10mg/dl (>= 100mg/l) and an abnormal serum free light chain ratio (< 0.26, or > 1.65)
  * Measurable biopsy proven plasmacytoma (should be measured within 28 days of initial investigational agent dosing)
* Patients must have had at least 2 prior line of therapy
* Patients must not have had progression of disease on lenalidomide 25 mg; stable disease on lenalidomide is permitted
* Patient may be enrolled at any time from last line of therapy
* Absolute neutrophil count (ANC) > 1000/uL
* Platelets >= 75,000/uL, if plasma cell percentage on bone marrow biopsy aspirate or core is > 30%, platelet eligibility requirement will be adjusted to 60,000/uL
* Total bilirubin =< 1.5 mg/dL
* Alkaline phosphatase =< 3 X the upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2 X the ULN
* Serum creatinine =< 2 mg/dL or calculated creatinine clearance of >= 40 ml/min within 14 days of registration using Modification of Diet in Renal Disease (MDRD) formula
* Patient must be able to swallow capsule or tablet
* Patients must provide informed consent
* Patients must have a left ventricular ejection fraction > 30%, no uncontrolled arrhythmias or New York Heart Association class III-IV heart failure
* Patients must have a Karnofsky performance status >= 70
* A negative pregnancy test will be required for all women of child bearing potential; breast feeding is not permitted
* Fertility requirements:

  * Female patients with child bearing potential must have a negative pregnancy test at least 7 days before starting treatment drugs
  * Male patients must agree to use an adequate method of contraception for the duration of the study and for 90 days afterwards
  * Female patients must be either posy-menopausal, free from menses >= 2 years (yrs), surgically sterilized, willing to use two adequate barrier methods of contraception to prevent pregnancy, or agree to abstain from sexual activity starting from screening and for 90 days afterwards
  * Female patients of child bearing potential must agree to comply with the fertility and pregnancy test requirements dictated by the Rev-Assist program

Exclusion Criteria:

* Patients with peripheral neuropathy > Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Prior exposure to anti programmed cell death 1 (PD1) or anti programmed cell death 1 ligand 1 (PDL1)
* Patients receiving concurrent corticosteroids at the time protocol therapy is initiated other than for physiologic maintenance treatment
* History of allergic reaction (including erythema nodosum) to lenalidomide
* Concurrent use of complementary or alternative medicines that would confound the interpretation of toxicities and antitumor activity of the study drugs
* Patients with contraindication to thromboprophylaxis
* Unacceptable cardiac risk factors defined by any of the following criteria: patients with congenital long QT syndrome, any history of ventricular fibrillation or torsade de pointes, bradycardia defined as heart rate (HR) < 50 bpm, left ventricular ejection fraction < 30%
* Patients who have received targeted or investigational agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies
* Patients who have undergone major surgery =< 2 weeks prior to starting study drug or who have not recovered from the side-effects of surgery
* Patients with known positivity for human immunodeficiency virus (HIV), or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention, other than non-melanoma skin cancer and carcinoma in situ of the cervix should not be enrolled; patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from a prior malignancy for >= 5 yrs and are considered by their physician to be less than 30% risk of relapse
* Patients with active (untreated or relapsed) central nervous system (CNS) metastasis of the patient's myeloma
* Patients with a history of gastrointestinal surgery or other procedure that might, in the opinion of the investigator(s), interfere with the absorption or swallowing of the study drugs
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to them by the study staff
* Any other medical condition, including mental illness or substance abuse, deemed by the investigator(s) to likely interfere with the patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
MTD of pidilizumab combined with lenalidomide defined as the dose level at which no more than one of 6 patients experiences a dose-limiting toxicity (Phase I) | 28 days
Overall response rate in responding patients according to the IMWG response criteria (Phase II) | Up to 30 days
  The proportion of responses (partial and complete) will be calculated out of all eligible patients who receive any treatment in that disease group who are included in the phase II assessment. Assuming the number of responses is binomially distributed, 95% binomial confidence intervals will also be calculated for the estimate of the proportion of responses.

SECONDARY OUTCOMES:
Time to progression | Time from start of treatment until progression or death, assessed up to 30 days
Overall survival (Phase II) | Time from start of treatment to the date of his or her death, assessed up to 30 days
  OS will be evaluated using the methods of Kaplan-Meier.
Pharmacokinetic parameters of pidilizumab in combination with lenalidomide | Baseline, immediately at the end of infusion, 1, 24, 72, 168, and 336 hours, and just prior to course 2

OTHER OUTCOMES:
Assess CT-011 Immunogenicity of pidilizumab | Up to 30 days
Assess Immunomonitoring of lymphoctes to includeT and NK cell subsets | Up to 30 days
  Extensive immunomonitoring of T and NK cell subsets at baseline and upon completion of each 28-d cycle of therapy will be conducted.
Ex-vivo assessment of immune functional activities | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Efebera, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT02077959/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT02077959/ICF_001.pdf